CLINICAL TRIAL: NCT05748353
Title: Endocrine Disruptors and Life STILe in Patients Carrying BRCA Pathogenic VAriants With Breast and/or Ovarian CAncer and Women Without Neoplasm: the STILVARCA Study
Brief Title: Endocrine Disruptors and Life STILe in Breast Cancer Development
Acronym: STILVARCA
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FABI ALESSANDRA, Principal Investigator, Director of Unit of Precision Medicine in Breast Cancer, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4472
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; BRCA1 Mutation; BRCA2 Mutation; Ovarian Cancer; Life Style; Cadmium Exposure
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with BRCA pathological variants with breast or ovarian cancers: Patient with pathogenetic mutation of BRCA 1 or 2 gene who have developed breast or ovarian neoplasm
- Patients with BRCA pathological variants without diagnosis of cancer: Patient with pathogenetic mutation of BRCA 1 or 2 gene without diagnosis of malignancy and without prophylactic surgery

SUMMARY:
The aim of the study is to evaluate the role of lifestyle and environmental factors ( environmental contaminants such as Cd) on the penetrance of BRCA1/2 genes in BRCAm patients with Breast cancer and/or Ovarian cancer and in BRCAm healthy women without cancer diagnosis

DETAILED DESCRIPTION:
Breast cancer (BC) is the most frequent neoplasm in women; the lifetime probability of developing invasive breast cancer is estimated to be 12.8%. Ovarian cancer (OC) represents the second most common type of gynecologic neoplasm, with an incidence of about 1.5%. A sedentary lifestyle and being overweight seem to play a role in the development of these diseases; an increase in body mass index (BMI) of 5 units is correlated with a 12% increased risk of developing BC and 7-10% increased risk of developing OC. Exposure to environmental toxic factors, such as Cadmium (Cd), has also been found to play a role in the development of BC and OC. Indeed, it has been shown that Cd is involved in the pathogenesis of these neoplasms as it would act as an endocrine disruptor: through binding to the estrogen receptor it would determine its activation thereby promoting cell proliferation. Cd is released into the soil, water and air from natural sources but, most importantly, as a result of industrial processing the processing of nonferrous metals, the production of batteries and paints, the production and application of phosphate-based artificial fertilizers, the use of coal and petroleum, incineration and waste disposal. The general population may be exposed to Cd through: contaminated food and drinking water; cigarette smoking (active and passive), as tobacco leaves accumulate Cd from the soil; and inhalation of dust and fumes, especially for people living near industries that process or emit Cd. At the same time, it is well known that genetic factors are also related to the pathogenesis of BC and OC. In about 20% of patients with triple-negative BC and 20-25% of women with high-grade serous OC, a pathogenetic variant of these genes can be found. In subjects carrying constitutional pathogenetic variants (VPs) in the BRCA1/2 (BRCA1/2m) genes, the absence of repair of damage to the DNA double helix causes its accumulation favoring the development of neoplasms. This results in individuals carrying these variants having a cumulative risk of developing BC of 72% in the case of BRCA1 and 62% in the case of BRCA2. With regard to OC, the risk associated with the presence of VP in the case of BRCA1 is 44% and 17% in the case of BRCA2. These observations are consistent with the hypothesis that genetic risk related to cancer development is modified by environmental or other molecular factors. Several studies have evaluated factors such as lifestyle, overweight, weight gain, and physical inactivity as potential risk elements of BC or OC in BRCA1/2m mutation carriers. The aim of this study is to evaluate the possible interference of environmental factors in the development of BC or OC in women VP carriers of BRCA 1 and BRCA 2

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Histologic diagnosis of early-stage BC (stage I, II, III operated; luminal, HER2+, triple-negative tumors) or OC (high-grade epithelial any stage and histotype); presence of germline variant of BRCA1 or BRCA2, class 4 or 5
* Patients carrying germline variant of BRCA1 or BRCA2, class 4 or 5, in the absence of BC and/or OC, who have not undergone prophylactic mastectomy and/or bilateral ovariectomy surgery.
* Patients with malignancy must have undergone surgery and be currently disease-free or in complete or partial remission in the case of OC.
* Adjuvant/neoadjuvant systemic therapy as well as maintenance therapy (PARP-inhibitors for example) is permitted.
* Signature of informed consent.
* ECOG: 0.1.
* Compliance with questionnaire completion

Exclusion Criteria:

* Prophylactic breast or ovarian surgery
* Germinal variant of BRCA1 or BRCA2, class 1,2, 3.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pathogenic mutation of BRCA1 or BRCA2 gene with/without development of BC and/or OC
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Adherence to mediterranean diet | 10 years
  Identification of adherence to the Mediterranean diet assessed through the PREDIMED questionnaire, a validated 14-item Questionnaire of Mediterranean diet adherence. The score can range from 0 to 14. A score less than 5 indicates poor adherence to the Mediterranean diet; a score between 6 and 9 means average adherence and greater than 10 good adherence.

SECONDARY OUTCOMES:
Assessment of fisical activity | 10 years
  Assessment of physical activity (assessed through the IPAQ questionnaire). Questionnaire measures the type and amount of physical activity performed by the subject during the week and it is divided into intense, moderate and light. Each activity is assigned a score. A total score below 700 Met indicates inactivity of the subject, between 701 and 2519 sufficient activity, above 2520 adequate activity
Assessment of smoke habits | 10 years
  An assessment of the subject's smoking habit. It evaluate the number of cigarettes smoked daily and years from beginning. The score is expressed by "pack-years" index.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, Principal Investigator — Medicina di precisione in senologia, policliclinico A. Gemelli - IRCCS
Locations (1):
- Alessandra Fabi, Roma, Italy